CLINICAL TRIAL: NCT05744804
Title: Efficacy and Safety of Low Dose Rivaroxaban in Patients With Anterior Myocardial Infarction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Mohamed Elamir Saber, resident doctor at internal medecine department, Sohag University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: soh-Med-23-01-09
Record Dates: First submitted 2023-02-16; First posted 2023-02-27 (Actual); Last update posted 2023-02-27 (Actual); Status verified 2023-02

CONDITIONS: Patient With Anterior Myocardial Infarction
MeSH Terms: interventions — Aspirin; Clopidogrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- -group of patients(75 patients) will receive low dose rivaroxaban (Active Comparator): -group of patients(75 patients) will receive low dose rivaroxaban (rivaroxaban 2.5 mg twice daily orally) for 1 month after anterior ST-segment myocardial infarction plus dual antiplatelet therapy (acetylsalicylic acid 75 mg once daily orally and cloppe
  Interventions: Drug: -group of patients(75 patients) will receive low dose rivaroxaban myocardial infarction plus (acetylsalicylic acid 75 mg and clopidogrel 75 mg
- control group of patients: (Active Comparator): control group of patients: 75 Patients of anterior ST-segment myocardial infarction on dual antiplatelet therapy only
  Interventions: Drug: (acetylsalicylic acid 75 mg once daily orally and clopidogrel 75 mg once daily orally only)

INTERVENTIONS:
Drug: -group of patients(75 patients) will receive low dose rivaroxaban myocardial infarction plus (acetylsalicylic acid 75 mg and clopidogrel 75 mg — receive low dose rivaroxaban (rivaroxaban 2.5 mg twice daily orally) for 1 month after anterior ST-segment myocardial infarction plus dual antiplatelet therapy (acetylsalicylic acid 75 mg once daily orally and clopidogrel 75 mg once daily orally)
  Arms: -group of patients(75 patients) will receive low dose rivaroxaban
Drug: (acetylsalicylic acid 75 mg once daily orally and clopidogrel 75 mg once daily orally only) — control group of patients: 75 Patients of anterior ST-segment myocardial infarction on dual antiplatelet therapy only
  Arms: control group of patients:

SUMMARY:
Despite the use of guideline directed optimal medical therapy, 12% of patients with stable coronary heart disease and 18% of patients with recent acute coronary syndrome experience recurrent major adverse cardiovascular events 1. The risk of recurrent cardiovascular events may be related to persistent elevation of thrombin beyond the index event 2,3

which leads to progression of cardiovascular disease by inducing inflammation, endothelial dysfunction and thrombosis 4. In patients with coronary heart disease, vitamin K antagonists (VKAs) and direct oral anticoagulants (DOACs) have been explored as secondary prevention strategies and have shown cardiovascular benefits at the cost of higher bleeding events 5,6,7,8.

howeverLeft ventricular thrombus (LVT) usually appearswithin 1 month after ST-segment elevation myocardial infarction (STEMI) and mostlyforms after anterior STEMI.9,11Although the prevalenceof LVT after acute myocardial infarction hasdecreased dramatically in modern times due to the progress of reperfusion therapy, LVT incidence in patients with anterior STEMI remains at 4% to 26%.10,12 It complicates acute myocardial infarction and is associated with a higher incidence of poor outcomes.9

ELIGIBILITY:
Inclusion Criteria:

* patients with anterior ST-segment myocardial infarction on acetylsalicylic acid and clopidogrel

Exclusion Criteria:

1. Patients with liver cirrhosis.
2. Patients with severe mitral stenosis .
3. Patients with bleeding tendency (HASBLED score ≥ 3)
4. Severe renal impairment ( creatinine clearance < 30 ml/min ).
5. patients with prosthetic valve .
6. patients on ticagrelor treatment
7. patients with Atrial Fibrillation

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 150 (Estimated)
Dates: Start 2023-03-01 (Estimated); Primary Completion 2023-12-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Major adverse cardiovascular event | 10 months
  Major adverse cardiovascular event
Left ventricular function | 10 months
  Left ventricular function
Left ventricular thrombus | 10 months
  Left ventricular thrombus
Transient Ischemic Attacks or cerebrovascular stroke | 10 months
  Transient Ischemic Attacks or cerebrovascular stroke

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bhatt DL, Eagle KA, Ohman EM, Hirsch AT, Goto S, Mahoney EM, Wilson PW, Alberts MJ, D'Agostino R, Liau CS, Mas JL, Rother J, Smith SC Jr, Salette G, Contant CF, Massaro JM, Steg PG; REACH Registry Investigators. Comparative determinants of 4-year cardiovascular event rates in stable outpatients at risk of or with atherothrombosis. JAMA. 2010 Sep 22;304(12):1350-7. doi: 10.1001/jama.2010.1322. Epub 2010 Aug 30. PMID 20805624
- [Background] Merlini PA, Bauer KA, Oltrona L, Ardissino D, Cattaneo M, Belli C, Mannucci PM, Rosenberg RD. Persistent activation of coagulation mechanism in unstable angina and myocardial infarction. Circulation. 1994 Jul;90(1):61-8. doi: 10.1161/01.cir.90.1.61. PMID 8026047
- [Background] Ueda Y, Ogasawara N, Matsuo K, Hirotani S, Kashiwase K, Hirata A, Nishio M, Nemoto T, Wada M, Masumura Y, Kashiyama T, Konishi S, Nakanishi H, Kobayashi Y, Akazawa Y, Kodama K. Acute coronary syndrome: insight from angioscopy. Circ J. 2010 Mar;74(3):411-7. doi: 10.1253/circj.cj-09-0795. Epub 2010 Jan 30. PMID 20118566
- [Background] Borissoff JI, Spronk HM, Heeneman S, ten Cate H. Is thrombin a key player in the 'coagulation-atherogenesis' maze? Cardiovasc Res. 2009 Jun 1;82(3):392-403. doi: 10.1093/cvr/cvp066. Epub 2009 Feb 19. PMID 19228706